CLINICAL TRIAL: NCT03489863
Title: Pharmacodynamic Comparison of Prasugrel Versus Ticagrelor in Patients With CYP2C19 Loss-of-function Genotype: a Validation Study in Patients With Stable Coronary Artery Disease
Brief Title: Prasugrel Versus Ticagrelor in Patients With CYP2C19 Loss-of-function: a Validation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Scott R. MacKenzie Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201703338 -A
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
Keywords: clopidogrel; prasugrel; ticagrelor
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prasugrel (Active Comparator): Patients will be randomly (1:1) assigned to receive FDA approved doses of either prasugrel (60 mg loading dose - 10 mg/day maintenance dose) or ticagrelor (180 mg loading dose - 90 mg b.i.d maintenance dose).
  Interventions: Drug: Prasugrel
- Ticagrelor (Active Comparator): Patients will be randomly (1:1) assigned to receive FDA approved doses of either prasugrel (60 mg loading dose - 10 mg/day maintenance dose) or ticagrelor (180 mg loading dose - 90 mg b.i.d maintenance dose).
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Maintenance dose will be maintained for 10±3 days.
  Other Names: Effient
  Arms: Prasugrel
Drug: Ticagrelor — Maintenance dose will be maintained for 10±3 days.
  Other Names: Brilinta
  Arms: Ticagrelor

SUMMARY:
Polymorphisms of the cytochrome P450 (CYP) 2C19 enzyme has been consistently shown to modulate clopidogrel response. Accordingly, the Food and Drug Administration (FDA) has issued a warning on the potential for reduced efficacy of clopidogrel among carriers of loss-of-function alleles (LOF) for CYP2C19 and suggest considering alternative antiplatelet therapies for these individuals.

The pharmacodynamic (PD) effects of prasugrel and ticagrelor are not affected by CYP2C19 genetic polymorphisms. However, to date there are no head-to-head PD comparisons between these agents among patients with different CYP2C19 genetic polymorphisms, which is currently under investigation in CAD patients undergoing PCI at UF Health-Jacksonville (UFJ 2014-12, NCT 02065479). In order to rule out play of chance findings, pharmacogenetic investigations require external validation cohorts to support the study findings. Therefore, the present randomized study is designed to serve as an external validation cohort conducted in patients with established CAD not undergoing PCI testing the non-inferiority in platelet reactivity of prasugrel versus ticagrelor among CYP2C19 LOF allele carriers.

DETAILED DESCRIPTION:
Therapeutic inhibition of platelet activation is essential for the management of ischemic cardiovascular disease. The use of platelet adenosine diphosphate (ADP) P2Y12 receptor antagonists (clopidogrel, prasugrel, and ticagrelor) in addition to aspirin are associated with a decrease in cardiovascular events in high-risk coronary artery disease (CAD) patients. Clopidogrel is the most broadly utilized P2Y12 receptor antagonist. However, among clopidogrel treated patients, there is broad variability in antiplatelet drug response which is known carry prognostic implications. Polymorphisms of the cytochrome P450 (CYP) 2C19 enzyme has been consistently shown to modulate clopidogrel response. Accordingly, the Food and Drug Administration (FDA) has issued a warning on the potential for reduced efficacy of clopidogrel among carriers of loss-of-function alleles (LOF) for CYP2C19 and suggest considering alternative antiplatelet therapies for these individuals.

The pharmacodynamic (PD) effects of prasugrel and ticagrelor are not affected by CYP2C19 genetic polymorphisms. However, to date there are no head-to-head PD comparisons between these agents among patients with different CYP2C19 genetic polymorphisms which is currently under investigation in CAD patients undergoing PCI at UF Health-Jacksonville (UFJ 2014-12, NCT 02065479). In order to rule out play of chance findings, pharmacogenetic investigations require external validation cohorts to support the study findings. Therefore, the present randomized study is designed to serve as an external validation cohort conducted in patients with established CAD not undergoing PCI testing the non-inferiority in platelet reactivity of prasugrel versus ticagrelor among CYP2C19 LOF allele carriers.

ELIGIBILITY:
Inclusion criteria:

* Patients with CAD [defined as the presence of at least a 50% stenosis in a major epicardial vessel or major branch, or any prior coronary revascularization (PCI or coronary bypass graft surgery)] on treatment with either aspirin (81mg/day) or aspirin and clopidogrel (75m/day) for at least 30 days as per standard of care
* Participated in UFJ 2016-14 study with genetic buccal swab test and have at least one CYP 2C19 LOF allele (CYP2C19*2 and CYP2C19*3)
* Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Exclusion criteria:

* Known allergies to prasugrel or ticagrelor
* Weight <60kg
* Considered at high risk for bleeding
* Currently active bleeding
* History of ischemic or hemorrhagic stroke or transient ischemic attack, or intracranial hemorrhage
* Known severe hepatic dysfunction
* On treatment with oral anticoagulant therapy (Vitamin K antagonists, dabigatran, apixaban, rivaroxaban)
* Platelet count <80x106/mL
* Hemoglobin <10 g/dL.
* Creatinine Clearance <30 mL/minute
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with ticagrelor): CYP3A Inhibitors (ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin ) and CYP3A Inducers (rifampin, phenytoin, carbamazepine, and phenobarbital)
* Pregnant or breastfeeding females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD,PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prasugrel | Ticagrelor
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Ticagrelor | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8) | 60 (8) | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
diabetes mellitus [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Unit (PRU)
Description: Platelet reactivity measured by VerifyNow and reported as PRU
Time Frame: at 24 hours post loading dose
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 7 | 6
PRU | 5 (10) | 24 (22)
Statistical Analysis 1: Comparison: Prasugrel vs Ticagrelor; The primary endpoint is non-inferiority in PRU, at 24 hours of prasugrel versus ticagrelor. Under the assumption of 0 difference at 24 hours in mean PRU between ticagrelor and prasugrel and a common standard deviation of 50 PRU, a sample size of 22 patients per group allows for the 95% CI to stay within ± 45 PRU with a 90% power and alpha = 0.05; Test type: Non-Inferiority — see above; p < 0.05, ANCOVA; Mean Difference (Net) = -18, 95% CI 2-sided [-38 to 2]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Prasugrel | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03489863/Prot_SAP_000.pdf